CLINICAL TRIAL: NCT06044402
Title: Effect of Intraoperative Low Tidal Volume vs Intermediate Tidal Volume on Oxygenation, Respiratory Mechanics, and Pulmonary Complications in Older Patients Undergoing Trendelenburg Pneumoperitoneum Surgery: A Randomized Clinical Trial
Brief Title: Different Tidal Volume on Oxygenation, Respiratory Mechanics, and Pulmonary Complications in Older Patients Undergoing Trendelenburg Pneumoperitoneum Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: dong zhang (Other)
Responsible Party: Sponsor-Investigator, dong zhang, Principal Investigator, Gansu Provincial Hospital
Organization: Gansu Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GanSu Province Hospital
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Trendelenburg; Neumoperitoneum; Oxygenation; Respiratory; Pulmonary

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group L (Placebo Comparator): Ventilation was subsequently changed to individualized positive end-expiratory pressure and recruitment maneuvers during trendelenburg pneumoperitoneum, and the tidal volume was set to 6 ml/kg.
  Interventions: Other: group L (Vt 6 ml/kg)
- group I (Experimental): Ventilation was subsequently changed to individualized positive end-expiratory pressure and recruitment maneuvers during trendelenburg pneumoperitoneum, and the tidal volume was set to 8 ml/kg.
  Interventions: Other: group I (Vt 8 ml/kg)

INTERVENTIONS:
Other: group L (Vt 6 ml/kg) — low tidal volume ventilation (tidal volume was set to 6 ml/kg)
  Arms: group L
Other: group I (Vt 8 ml/kg) — intermediate tidal volume ventilation (tidal volume was set to 8 ml/kg)
  Arms: group I

SUMMARY:
The investigators want to assess the effect of intraoperative low tidal volume vs intermediate tidal volume on respiratory mechanics, oxygenation and pulmonary complications in older patients undergoing Trendelenburg pneumoperitoneum surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III class;
* Colorectal cancer patients;
* Elective laparoscopic colorectal surgery;
* expected duration of surgery greater than 2 hours.

Exclusion Criteria:

* serious complications associated with other systems;
* severe cardiac insufficiency;
* renal failure;
* body mass index (BMI) greater than 30 kg/m2 or less than 18 kg/m2;
* the use of low tidal volume and consequent hypercapnia can induce harm;
* refusal to participate in the study.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 | the lowest value at one hour after extubation, day-1 to day-3
  the outcome in mmHg
hypoxemia | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
pneumonia | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
bronchospasm | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
atelectasis | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
pulmonary congestion | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
respiratory failure | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
pleural effusion | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
pneumothorax | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction
unplanned requirement for postoperative invasive or noninvasive ventilation | From date of patient admission until the date of discharge, assessed up to 7 days
  the outcome in fraction

SECONDARY OUTCOMES:
Tidal volume | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in milliliter
respiratory rate | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in times/minute (frequency)
dead space fraction | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in fraction
A-aDO2 | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in mmHg
intrapulmonary shunt | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in fraction
peak airway pressure | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in cmH2O
plateau airway pressure | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in cmH2O
mean airway pressure | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in cmH2O
dynamic compliance | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3)
  the outcome in milliliter/cmH2O
arterial blood pH | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in number
arterial blood PO2 | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmHg
arterial blood PCO2 | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmHg
arterial blood Hb | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in g/dl
arterial blood Hct | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in fraction
arterial blood SO2 | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in fraction
arterial blood K | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood Na | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood Ca | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood Cl | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood Glu | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood Lac | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood tBil | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in umol/L
arterial blood SBE | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
arterial blood ABE | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmol/L
PaO2/FiO2 | before anesthesia induction (T1); 60 minutes after initiation of the Trendelenburg position and CO2 pneumoperitoneum (T2), and 10 minutes after desufflation and resuming the supine position (T3).
  the outcome in mmHg
unplanned intensive care unit admission | From date of finishing surgery until the date of patient discharge, assessed up to 7 days
  the outcome in fraction
intensive care unit length of stay | From date of finishing surgery until the date of patient discharge, assessed up to 7 days
  the outcome in days
postoperative mortality | From date of finishing surgery until the date of patient discharge, assessed up to 7 days
  the outcome in fraction
hospital length of stay | From date of patient admission until the date of discharge, assessed up to 10 days
  the outcome in days